CLINICAL TRIAL: NCT05007444
Title: Determination of the Optimal Biological Dose and Safety Evaluation of the P2Et Extract in Patients With Breast Cancer (Phase I / II)
Brief Title: Safety and Efficacy Evaluation of the P2Et Extract in Patients With Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS003-BC
Record Dates: First submitted 2021-08-02; First posted 2021-08-16 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Quality of Life; Tumor, Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a design based on adaptive randomized simulations (BOIN12) (Zhou, Lee, & Yuan, 2019). Each of the patients included in the different groups will undergo the analysis of the immune response parameters described in Annex 1.
  With the optimal biological dose calculated in stage 1, it will go to stage 2 where 40 randomized breast cancer patients will be enrolled in treatment with the P2Et extract or placebo. In these patients, parameters related to the immune response, progression-free survival, quality of life and tumor reduction will be evaluated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo comparator (Placebo Comparator): Patients in the placebo group will receive the stable daily dose divided into 2 doses with meals of the optimal biological dose determined in stage I every 12 hours for the duration of standard therapy. The patient will self-administer the phytomedicine until completing the established treatment days. The taking of the phytomedicine will only be suspended 3 days before each cycle of standard therapy and will restart 3 days after having passed the cycle. That is, in the anthracycline and cyclophosphamide (AC) phase, the patient will start taking the phytomedicine 3 days after having received their standard chemotherapy cycle and will suspend it 3 days before the next cycle begins. For the taxane phase, the patient will take the P2Et without suspension during the treatment cycles.
  Interventions: Drug: Placebo
- Active comparator P2Et (Active Comparator): Patients in the P2Et group will receive the stable daily dose divided into 2 doses with meals of the optimal biological dose determined in stage I every 12 hours for the duration of standard therapy. The patient will self-administer the phytomedicine until completing the established treatment days. The taking of the phytomedicine will only be suspended 3 days before each cycle of standard therapy and will restart 3 days after having passed the cycle. That is, in the anthracycline and cyclophosphamide (AC) phase, the patient will start taking the phytomedicine 3 days after having received their standard chemotherapy cycle and will suspend it 3 days before the next cycle begins. For the taxane phase, the patient will take the P2Et without suspension during the treatment cycles.
  Interventions: Drug: P2Et (Caesalpinia spinosa extract)

INTERVENTIONS:
Drug: P2Et (Caesalpinia spinosa extract) — Patients who meet inclusion criteria will begin taking 4000mg daily, distributed in 2 doses with meals of 2000mg of P2Et extract during neoadjuvant treatment. In case of presenting toxicity, it will be lowered to the next dose level, that is, 2000 mg under the same dosage schedule and 1000 mg following the same principle. The taking of the phytomedicine will only be suspended 3 days before each cycle of standard neoadjuvant therapy and will restart 3 days after having passed the cycle. That is, in the anthracyclines and cyclophosphamide (AC) phase, the patient will start taking the phytomedicine 3 days after having received their standard chemotherapy cycle and will suspend it 3 days after the next cycle begins. For the taxane phase, the patient will take the P2Et without suspension during the treatment cycles.
  Arms: Active comparator P2Et
Drug: Placebo — After determining the optimal biological dose (OBD), the patients will be divided into the placebo arm or the treatment arm. In the anthracyclines and cyclophosphamide (AC) phase, the patient will start taking according to the asignation as stated in the drug intervention.
  Arms: Placebo comparator

SUMMARY:
Currently, the study of many extracts in different types of cancer has allowed the validation of scientific knowledge either as a therapy that reduces the size of the tumor or that helps to improve the quality of life of the patient by reducing the associated effects of the treatment.

In the Immunobiology and Cell Biology group of the Pontificia Universidad Javeriana, a standardized extract of Caesalpinia spinosa (Dividivi) called P2Et has been obtained. This extract has been shown to have cytotoxic activity in different human and murine tumor cell lines, favoring the induction of immunogenic cell death with the release of danger signals such as calreticulin, HMGB1 and ATP. Additionally, treating mice with murine melanoma and sinus tumors significantly reduces tumor size and metastases. On the other hand, induction of complete autophagic flux and synergistic effects with anthracycline-type chemotherapeutics have been shown in human cell lines and in animal models of breast cancer.

With this background, and the results of the Phase I clinical study carried out in healthy volunteers that showed that the extract is safe, the investigators propose that treatment with the P2Et extract in patients with breast cancer could improve their general condition, impacting their quality of life. , and induce antitumor immune response, improving the immune infiltrate and acting as a transforming agent from a cold tumor to a warm tumor. This would lead to an improvement in the long-term survival of patients treated with the phytomedicine in conjunction with the chemotherapeutic treatment selected by the treating oncologist.

In order to advance on this path, and responding to the adjustments suggested in the phase I study in healthy individuals, it is proposed to carry out a clinical study that allows determining the optimal biological dose of the P2Et extract in a design based on randomized simulations of adaptive form and considering the safety of the extract as an objective in patients with breast cancer. Additionally, those parameters that allow defining the best indicators of effectiveness of P2Et in this group of patients will be evaluated, such as modulation of the immune response, quality of life, reduction of adverse effects and progression-free survival.

DETAILED DESCRIPTION:
Natural products and traditional herbal medicine are an important source of alternative bioactive compounds, but very few herbal preparations have been scientifically evaluated and validated for their potential as treatments in medical practice. Phytotherapy is a promising field in current therapies based on plant-derived compounds given its immunomodulation properties and its ability to act against tumors, favoring the activation of the immune response and the reversal of the tumor phenotype through its action on the tumor microenvironment.

Over the last 8 years, the investigators have shown that a standardized extract of Caesalpinia spinosa, which the investigators call P2Et and which is the study drug of this protocol, presents an antioxidant activity both intracellular and in solution, which is much higher than that of of the positive controls used as the TROLOX. P2Et can also modulate drug resistance pumps, increasing sensitivity to anthracyclines in vitro and in vivo. It induces apoptosis through the depolarization of the mitochondria in various tumor cells and specifically in murine breast cancer cells, decreases clonogenicity, which seems to be related to the reduction of the primary tumor and metastases in animal models of breast cancer. It can also decrease the production of serum IL-6 in these animals, possibly related to a reduction in the protumorigenic activity of tumor-associated fibroblasts (results not yet published). The P2Et-induced tumor death process is accompanied by the expression of immunogenic death markers such as the expression of calreticulin, secretion of HMGB1 and ATP, which participate in the activation of dendritic cells. Vaccination of the animals with tumor cells treated with P2Et allows the generation of long-lived memory LTs, producers of IFN-gamma, TNF-alpha and IL-2, 4 and 5, which can be detected ex vivo. In vivo in animals, treatment with a vaccine prepared with tumor cells treated with P2Et favors the recruitment and differentiation of LT to the draining lymph nodes, which produce cytokines in response to tumor antigens, showing their ability to recognize the tumor. The investigators were also able to show that P2Et induces a tumor-specific immune response that is superior to that induced by Doxorubicin, since the LTs generated present greater multifunctionality in terms of cytokine production. Doxorubicin is known to also induce an immune response through immunogenic cell death, however, it has also been observed that treatment with anthracyclines can favor the selection of CMT within the tumor, which suggests that although they induce antitumor immune response, it is necessary to improve the recognition of MTCs by the immune system. Vaccination of animals with wild type 4T1 tumor cells treated with P2Et can induce cytotoxic LTs capable of recognizing murine 4T1 tumor MTCs called H17. This strongly suggests that there are cross-reactive antigens in both tumor lines and that in vivo, treatment with P2Et could induce a cross-presentation of antigens that allows the activation of CMT-specific LTs, which would be reflected in a greater disease-free survival. in animals, and that the same could be observed in patients.

The ability of P2Et to carry out its antitumor activity has also been observed in a murine model of melanoma, in which the investigators show that treatment with P2Et induces LT CD8 specific for the melanoma-specific tumor antigen Trp-2, through a effective cross-presentation and antigenic presentation by dendritic cells. In fact, the antitumor activity of P2Et was reduced in RAGg KO immunodeficient animals, which do not present LT or LB, confirming that the effect of this phytomedicine is partially mediated by the immune response and that the immune response is required to be activated, to exercise its function.

The antitumor activity of P2Et may be due to the particular form of immunogenic cell death induction that is different from that induced by anthracyclines, which allows tumor antigens to not easily degrade when the cell is dying, due to its high capacity. antioxidant, which is concomitant with the expression by the tumor cell of immunogenic cell death markers. These two elements, together, allow dendritic cells to carry out better antigen processing with complete antigens and therefore the diversity of the LT response, measured at the clonotypic level, is greater.

The investigators are currently evaluating the local intratumoral and peripheral immune response induced by anthracycline treatment in patients with breast cancer at Hospital San Ignacio, in conjunction with a clonotypic analysis of the LTs generated in both compartments (unpublished data). These results will serve as a basis for later comparing whether the quality of the response in patients treated with P2Et in conjunction with conventional chemotherapy is different and whether this may be related to its antitumor activity in vivo.

On the other hand, in previous studies it has been observed that P2Et can modulate the expression of PD-L1 in tumor cells, improving the therapeutic effect of the anti PD-L1 antibody in vivo in a murine melanoma model. Although the same additive response to co-treatment (P2Et + anti-PD-L1) was not observed in the breast cancer model, protection of the affected hematopoietic cells was evidenced with anti-PD-L1 therapy with an improvement in the number of platelets, lymphocytes, monocytes and granulocytes in animals that received P2Et in conjunction with anti-PD-L1 compared to those that only received anti-PD-L1. The differences in melanoma and breast could be due to the increase in the expression of PD-L1 mainly in the murine melanoma line and not in the 4T1 line in response to P2Et, so it is important to measure the effect of the P2Et extract on the PD-L1 expression in human tumor cells and study the relationship with tumor type and other biological variables.

With this background, and the results of the Phase I clinical study carried out in healthy volunteers that showed that the extract is safe, the investigators propose that treatment with the P2Et extract in patients with breast cancer could improve their general condition, impacting their quality of life. , and induce an antitumor immune response, improving the immune infiltrate and acting as a transforming agent from a cold tumor to a warm tumor. This would lead to an improvement in the long-term survival of patients treated with phytomedicine in conjunction with the chemotherapeutic treatment selected by the treating oncologist.

In order to advance on this path, and responding to the adjustments suggested in the phase I study in healthy individuals, it is proposed to carry out a clinical study that allows determining the optimal biological dose of the P2Et extract in a design based on randomized simulations of adaptive form and considering the safety of the extract as an objective in patients with breast cancer. Additionally, those parameters that allow defining the best indicators of the effectiveness of P2Et in this group of patients will be evaluated, such as modulation of the immune response, quality of life, reduction of adverse effects and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women over 18 years of age.
2. Patients with a diagnosis of histopathologically confirmed stage II-III invasive breast cancer who are candidates for treatment with standard neoadjuvant chemotherapy.
3. Documented results of the status of estrogen receptors (ER), progesterone (RP), KI 67, and epidermal growth factor receptor 2 (HER-2).
4. Patients eligible for neoadjuvant treatment with AC (Doxorubicin / cyclophosphamide) every 2 or 3 weeks followed by taxanes (paclitaxel for 12 weeks or docetaxel every 3 weeks for 4 cycles)
5. ECOG scale status from 0 to 1 with survival greater than 3 months.
6. Subject is able to swallow and retain oral medication and does not have uncontrolled emesis or persistent diarrhea.
7. Adequate renal, hematological, and hepatic function at the discretion of the investigator.
8. No uncontrolled or significant comorbidities determined by medical history, physical examination and screening laboratories at the discretion of the investigator. (Leukocytes greater than 2000 / mm3, neutrophils greater than 1500 / mm3, hemoglobin greater than 9 g / dl, creatinine less than 1.5 times the upper limit, transaminases less than 3 times the upper limit, bilirubin less than 1.5 times the upper limit).
9. Patients of childbearing age and without safe non-hormonal planning methods should have a negative pregnancy test before screening and each treatment cycle.
10. Fertile female subjects (those who are not postmenopausal for at least 12 months or are surgically sterile by bilateral tubal ligation, bilateral oophorectomy or hysterectomy) and their male partners, must use at least one of the contraceptive methods that are listed below during study entry, throughout the study, and for at least 6 months after use of the P2Et extract (the effects of the P2Et extract on the developing human fetus are unknown):

to. Complete abstinence from sexual intercourse, beginning at least one complete menstrual cycle before administration of study drug; (It should be noted: sexual abstinence as a contraceptive method should be limited to those cases in which it is already established as the choice of the patient's pre-existing lifestyle).

b. Vasectomy in the partner of a female subject c. Intrauterine device (IUD) d. Double barrier method (condom, contraceptive sponge, diaphragm or vaginal ring with jelly or spermicidal cream).

k) Desire to complete the study and follow-up interventions.

Exclusion Criteria:

1. Subjects treated in any other clinical therapeutic protocol in the 30 days prior to study entry or during study participation.
2. Patients who are receiving other agents under investigation.
3. History of allergic reactions attributed to polyphenol-type compounds similar to those found in green tea.
4. The subject is a pregnant or breastfeeding woman.
5. Patients who due to their clinical condition should receive anti-HER2 antibodies
6. Concomitant severe morbidity, active at the discretion of the investigator
7. Subjects with malabsorption syndrome or another condition that affects the enteral route of administration
8. Subjects with confirmed HIV diagnosis prior to enrollment or HIV positive diagnosis at the time of screening.
9. Solid organ transplant recipients or hematopoietic component.
10. The use of other phytomedicines, vitamins or herbal supplements must have been suspended at least one week before entering the study.
11. Previous malignant disease active within the previous 3 years, except for locally curable cancers that have apparently been cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix or mother
12. Any condition that at the discretion of the principal investigator renders the subject ineligible to participate in this study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Toxicological profile | 18 months
  Determination of the optimal Biological Dose according to the toxicological profile

SECONDARY OUTCOMES:
Clinical and pathological response in the tumor of the patients | 18 months
  To determine the effect of treatment with P2Et extract and neoadjuvant chemotherapy on the clinical and pathological response in the cohort.
Survival | 24 months
  To assess the disease-free survival of breast cancer patients treated with the P2Et extract in the expanded cohort of patients.
Quality of life in breast cancer patients | 24 months
  To evaluate the effect of treatment with P2Et extract and neoadjuvant chemotherapy on the quality of life of patients with breast cancer by applying the QLQ C-30 version 3 questionnaire and QLQ B23 in the expanded cohort of
Adverse events | 18 months
  Evaluate the adverse events of the P2Et extract in combination with neoadjuvant chemotherapy in breast cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Bardia A, Baselga J. Neoadjuvant therapy as a platform for drug development and approval in breast cancer. Clin Cancer Res. 2013 Dec 1;19(23):6360-70. doi: 10.1158/1078-0432.CCR-13-0916. PMID 24298066
- [Background] Bayet-Robert M, Kwiatkowski F, Leheurteur M, Gachon F, Planchat E, Abrial C, Mouret-Reynier MA, Durando X, Barthomeuf C, Chollet P. Phase I dose escalation trial of docetaxel plus curcumin in patients with advanced and metastatic breast cancer. Cancer Biol Ther. 2010 Jan;9(1):8-14. doi: 10.4161/cbt.9.1.10392. Epub 2010 Jan 21. PMID 19901561
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Burnet FM. The concept of immunological surveillance. Prog Exp Tumor Res. 1970;13:1-27. doi: 10.1159/000386035. No abstract available. PMID 4921480
- [Result] Ali HR, Provenzano E, Dawson SJ, Blows FM, Liu B, Shah M, Earl HM, Poole CJ, Hiller L, Dunn JA, Bowden SJ, Twelves C, Bartlett JM, Mahmoud SM, Rakha E, Ellis IO, Liu S, Gao D, Nielsen TO, Pharoah PD, Caldas C. Association between CD8+ T-cell infiltration and breast cancer survival in 12,439 patients. Ann Oncol. 2014 Aug;25(8):1536-43. doi: 10.1093/annonc/mdu191. Epub 2014 Jun 9. PMID 24915873
- [Derived] Ballesteros-Ramirez R, Pinilla P, Sanchez J, Torregrosa L, Aschner P, Uruena C, Fiorentino S. Safety and efficacy of P2Et extract from Caesalpinia spinosa in breast cancer patients: study protocol for a randomized double blind phase II clinical trial (CS003-BC). BMC Complement Med Ther. 2023 Sep 5;23(1):309. doi: 10.1186/s12906-023-04139-w. PMID 37670337